CLINICAL TRIAL: NCT04892407
Title: A Prospective, Multi-center, Randomized, Controlled, Single-blind Study of the Safety and Effectiveness of Algeness® DF 3.5% Deep Volumizing Filler to Correct Age-related Volume Deficit in the Mid-face
Brief Title: Algeness DF 3.5% Compared to Voluma in Volume Deficit in Mid-face
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Advanced Aesthetic Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AG35MF001
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Age-Related Volume Deficit in the Mid-Face

STUDY DESIGN:
Intervention Model Description: 3:1 randomization to either study product or comparator. If subject loses volume in cheek and/or returns to baseline score at or after 12month visit, he/she may be treated with study product.
Who Masked: Participant, Outcomes Assessor
Masking Description: The evaluator is blinded as to patient treatment. Patients are also not told what treatment they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Algeness DF 3.5% (Experimental): This arm is with the Sponsor's product. The product is already CE Marked and sold for this indication for the majority of participating countries.
  Interventions: Device: Algeness® DF 3.5%
- Juvéderm Voluma (Active Comparator): This arm is with a Control product that is already CE Marked and sold for this indication.
  Interventions: Device: Juvéderm Voluma

INTERVENTIONS:
Device: Algeness® DF 3.5% — dermal filler CE Mark approved for treatment of cheek and midface volume loss
  Arms: Algeness DF 3.5%
Device: Juvéderm Voluma — dermal filler CE Mark approved for treatment of cheek and midface volume loss
  Arms: Juvéderm Voluma

SUMMARY:
A prospective, randomized, controlled study of Algeness® DF 3.5% Deep Volumizing Filler comparing to Juvéderm Voluma to correct midface volume loss.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 22 years of age.
2. Subject has moderate to severe age-related volume deficit in the midface on both sides of the face as rated on LifeSprout Midface Scale, a proprietary, validated mid-face volume deficit scale
3. Subject willing to abstain from other facial aesthetic procedures in the mid-face through the last study follow-up visit which could interfere with treatment outcomes (e.g., facial fillers, skin laser and radiofrequency therapy such as Thermage, chemical re-surfacing, dermabrasion, Botox injections, aesthetic facial surgery, other facial treatments of the mid-face).
4. Subject willing and able to comply with study follow-up procedures and schedule.
5. Subject willing to provide written informed consent for their participation in the study.

Exclusion Criteria:

1. Subject is a female of childbearing potential (e.g., not postmenopausal for at least one year or has not had a hysterectomy or tubal ligation) not using medically effective birth control (e.g., hormonal methods in use at least 30 days prior to injection or barrier methods such as condom and spermicide in use at least 14 days prior to injection) or is pregnant, lactating, or plans to become pregnant during the study.
2. Subject has participated in a clinical study in which an investigational device or drug was received in the 30 days prior to screening or plans to enroll in such a study during the course of the current study.
3. Subject is an employee or direct relative of an employee of the investigational site or Sponsor.
4. Subject who has received surgery in the mid-face (including mesh, or threads), or has plans to during the study.
5. Subject has a serious or progressive disease, which, in the investigator's judgment, put the subject at undue risk (e.g., uncontrolled diabetes, autoimmune pathology, cardiac pathologies).
6. Subject has an acute inflammatory process or infection, or history of chronic or recurrent infection or inflammation with the potential to interfere with the study results or increase the risk of adverse events.
7. Subject has a disorder that may impact wound healing such as connective tissue or immunosuppressive disorder.
8. Subject has a history of precancerous lesions/skin malignancies.
9. Subject has had an active skin disease within the past 6 months.
10. Subject has scars, infection, rosacea, herpes, acne, blotches or other pathology on the mid-face.
11. Subject has facial hair in the mid-face that they are unwilling to remove for study assessments.
12. Subject is predisposed to keloidosis or hypertrophic scarring.
13. Subject has a known history of hyper- or hypo-pigmentation in the mid-face.
14. Subject has known allergy to agarose gel, algae, phosphate buffered saline, hyaluronic acid, gram positive bacterial proteins, streptococcal protein or lidocaine.
15. Subject has a known bleeding disorder.
16. Subject has received within the past week or plans to receive with 1 week before or up to 1 month after any treatment high-dose Vitamin E, aspirin, anti-inflammatories, antiplatelets, thrombolytics, or any other medication that could increase the risk of bleeding.
17. Subject has received within the past 3 months or plans to receive during the study chemotherapy agents, immunosuppressive medications, or systemic corticosteroids (inhaled steroids are acceptable).
18. Subject has received within the past 12 months or plans to receive during the study any injections outside of those in the study protocol including non-permanent fillers (e.g., hyaluronic acid, CaHA)
19. Subject has received within the past 12 months or plans to receive during the study neurotoxin on the face below the orbital rim (forehead is acceptable).
20. Subject has received at any time or plans to receive during the study a permanent filler (e.g., polylactic acid, PMMA, silicone) on the face.
21. Subject has received within the past 6 months or plans to receive during the study dermal resurfacing procedures or non-invasive skin tightening on the face.
22. Subject has received in the past 4 weeks or plans to receive during the study prescription facial wrinkle therapies (RENOVA), topical steroids, skin irritating topical preparations, or self-tanning agents on the face.
23. Subject has a known history of or plans during the study rapid weight loss/gain (5% of body weight).

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
with ≥ 1 point improvement from baseline on Proprietary Midface Scale, a validated midface volume deficit scale as rated by a live, masked evaluator | 6 month
  Statistical non inferiority of Study Product to Control by live Masked Evaluator of Subjects showing atleast a 1 point improvement. LifeSprout Midface Scale (0-4 with 0 being best and 4 being the worst/most extreme)

SECONDARY OUTCOMES:
1+ grade Improvement on Midface Scale Live Masked Evaluator All timepoints | 1, 3, 9, 12, 18, 24 months
  1+ grade improvement from baseline in midface scale by masked evaluator. LifeSprout Midface Scale (0-4 with 0 being best and 4 being the worst/most extreme)

OTHER OUTCOMES:
Change From Baseline Midface Scale Live Masked Evaluator All timepoints | 1, 3, 9, 12, 18, 24 months
  Individual endpoints for change from baseline on the Midface Scale as rated by a live, masked evaluator. LifeSprout Midface Scale (0-4 with 0 being best and 4 being the worst/most extreme)
GAIS Live Masked Evaluator | 1, 3, 9, 12, 18, 24 months
  GAIS Scores of Study Product and Comparator on Global Aesthetics Improvement Scale (GAIS) by live Masked Evaluator
GAIS Investigator | 1, 3, 9, 12, 18, 24 months
  GAIS Scores of Study Product and Comparator on Global Aesthetic Improvement Scale (GAIS) by Treating Investigator
GAIS Patient | 1, 3, 9, 12, 18, 24 months
  GAIS Scores of Study Product and Comparator on Global Aesthetic Improvement Scale (GAIS) by Patient
Patient Reported FACE-Q | 1, 3, 9, 12, 18, 24 months
  FACE-Q Satisfaction with Cheeks and Age Appraisal scales
Treatment Duration | 1, 3, 6, 9, 12, 18, 24 months
  Duration of treatment effect as measured on the Midface Scale by ≥1 point improvement, for those subjects who did not receive retreatment prior to the assessment timepoint at months 18 and 24.
Midface Photo | 1, 3, 6, 9, 12, 18, 24 months
  treatment effect as measured on the Midface Scale by ≥1 point improvement as graded by a blinded photographic reviewer
Midface Photo Change from Baseline | 1, 3, 6, 9, 12, 18, 24 months
  Individual endpoint of change from baseline score on the Midface Scale as rated by blinded photographic reviewer

CONTACTS AND LOCATIONS:
Locations (9):
- J. Vandeputte, Plastische Chirurgie, Oudenaarde, Belgium
- France (2):
  - MEDITI, Antibes
  - THINKIN, Paris
- Germany (2):
  - Rosenpark Research GmbH, Darmstadt
  - Private Practice for Dermatology and Aesthetics, Munich
- Shamir Medical Center, Ẕerifin, Israel
- Clique Clinic, Petaling Jaya, Malaysia
- Beauty Beyond Skin (Ocean Clinic Marbella), Marbella, Spain
- Galadari Derma Clinic, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
All summary results will be posted to this website. Safety results will be shared with medical monitor and study physicians.